CLINICAL TRIAL: NCT06571435
Title: Relationship Between Modified Closed Kinetic Chain Upper Extremity Stability Test and Shoulder Endurance Test in Young Active and Sedentary Individuals
Status: Recruiting | Type: Observational
Sponsor: Acibadem University (Other)
Collaborators: Biruni University (Other)
Responsible Party: Sponsor
Other Study IDs: AcibademU/2024-1/21
Record Dates: First submitted 2024-08-14; First posted 2024-08-26 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: endurance; shoulder; stability; young adult; sedentary
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active young adult: Participants will be assess with International Physical Activity Questionnaire(IPAQ-SF), which measures the duration of vigorous and moderate activity, walking and sitting over the previous 7 days. After they are done with the questionnaire, if they have >3000 MET/week score they will be considered as highly active group.
  Interventions: Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST), and Posterior Shoulder Endurance Test
- Sedentary young adult: Participants will be assess with International Physical Activity Questionnaire(IPAQ-SF), which measures the duration of vigorous and moderate activity, walking and sitting over the previous 7 days. After they are done with the questionnaire, if they have <600 MET/week score they will be considered as sedentary group.
  Interventions: Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST), and Posterior Shoulder Endurance Test

INTERVENTIONS:
Diagnostic Test: Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST), and Posterior Shoulder Endurance Test — The modified closed kinetic chain upper extremity stability test is reliable and is performed in an individualized manner by placing the hands on the floor at shoulder level. The evaluation process is the same as the original test; the total number of touches in 15 seconds is noted by lifting one hand, touching the other and placing it back. A total of 3 measurements are taken with a 45-second rest interval. The endurance capacity of the muscle group is an important factor for sports performance as it requires specific sports movements repeated in a certain period of time.
  For posterior shoulder endurance test participants will lie with their face down. While the shoulder is hanging from the stretcher, individuals will be asked to lift the dumble calculated with the weight appropriate for their weight to 90 degrees abduction in accordance with the 60 bpm metronome. Their duration in seconds will be noted. 1 measurement will be made with each arm.

SUMMARY:
This study is planned to examine the relationship between Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) performance with Posterior Shoulder Endurance Test in healthy young adults. Both tests are frequently used in athletes, but their use in sedentary people is not common in the literature. The feasibility of using these tests in sedentary people is not clear.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults aged between 18-25
* Volunteered for the study

Exclusion Criteria:

* Participants who had any injury on upper extremity in last 6 months
* Participants with moderately active results on IPAQ-SF

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young adults aged between 18-25 years old
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-08-14 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Closed Kinetic Chain Upper Extremity Stability Test (CKCUEST) Performance | 4 weeks
  Within 15 seconds, the total number of touches is noted. A total of 3 measurements are taken with a 45-second rest break
Posterior Shoulder Endurance Test Performance | 4 weeks
  Participants will lie face down. While the shoulder is hanging from the stretcher, individuals will be asked to lift the dumble calculated with the weight appropriate for their weight to 90 degrees abduction in accordance with the 60 bpm metronome. The time they can continue will be noted. 1 measurement will be made with each arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Acibadem University, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided